CLINICAL TRIAL: NCT04190680
Title: Kokkerelli Learning Street Effect Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20191129
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2023-09

CONDITIONS: Fruit and Vegetable Consumption in Children
Keywords: Nutrition; Fruit and vegetables; School; Children; Prevention

STUDY DESIGN:
Intervention Model Description: The study will consist of one intervention group (several primary school classes that participate in the Kokkerelli Learning Street) and one control group (several primary school classes that don't participate in the Kokkerelli Learning Street and continue with their regular curriculum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kokkerelli Learning Street (Experimental): The classes included in this group will participate in the Kokkerelli Learning Street; a school-based nutrition education programme included classroom-based lessons, a visit to a grower's farm and a cooking workshop.
  Interventions: Behavioral: Kokkerelli Learning Street
- Control group (No Intervention): The classes included in this group will not participate in the Kokkerelli Learning Street and will continue with their regular curriculum.

INTERVENTIONS:
Behavioral: Kokkerelli Learning Street — The Kokkerelli Learning Street focusses on one specific food product (kale, tomato, asparagus, pepper, strawberry, blue berry, mushroom, carrot, or leek) and consists of multiple components:
  1. An introduction lesson at school. Children are introduced to the product and familiarised with growing and harvesting processes and the importance of the product regarding health.
  2. A visit to a grower's farm during which children are introduced to the precise planting, growing and harvesting procedures of the product. Children are allowed to enter the facilities (e.g., the greenhouse) and observe and experience the farming of the product.
  3. A cooking workshop at the facilities of Kids University for Cooking BV. Children prepare a meal with help of volunteers. After preparing the meal, children help to set the table and consume their self-prepared meal.
  4. An evaluation lesson at school. Children evaluate the Learning Street together with their peers and teacher.
  Arms: Kokkerelli Learning Street

SUMMARY:
In 2012, the Kids University for Cooking Foundation BV has developed a nutrition education programme called 'Kokkerelli Learning Street'. This innovative programme aims to teach primary school students from study years 5-8 where food comes from, how it is processed, and how it can be used for the preparation of a healthy meal.

The Kokkerelli Learning Street is offered to primary school children in the region of Venlo, the Netherlands. The present study will investigate the effects of the Kokkerelli Learning Street on several determinants of children's fruit and vegetable intake. Based on the literature and the aims of the Learning Street, five relevant determinants are selected: (i) knowledge; (ii) taste preferences; (iii) intention; (iv) skills; and (v) attitude.

Using child-reported questionnaires, the present study aims to answer the following key questions:

What are the short-term and longer-term effects of the Kokkerelli Learning Street on children's:

* Knowledge regarding fruit and vegetable consumption?
* Intentions regarding fruit and vegetable consumption?
* Attitude regarding fruit and vegetable consumption?
* Liking of fruit and vegetables?
* Skills regarding fruit and vegetable preparation?
* Fruit and vegetable intake?

DETAILED DESCRIPTION:
In 2012, the Kids University for Cooking Foundation BV has developed a nutrition education programme called 'Kokkerelli Learning Street'. This innovative programme aims to teach primary school students aged 8-12 years (study years 5-8) where food comes from, how it is processed, and how it can be used for the preparation of a healthy meal. The theoretical foundation of the Learning Street is based on the EnRG framework, which states that behaviour is influenced both by conscious and unconscious processes. These processes can (in)directly be influenced by environmental factors. In addition, several behavioural and personal factors are thought to moderate the causal path.

The Kokkerelli Learning Street is offered to primary school children in the region of Venlo, the Netherlands. It involves education based on concepts of the Self-Determination Theory, active learning, and imagineering (e.g., self-experience in an interactive environment, rather than conventional education). The present study will investigate the effects of the Kokkerelli Learning Street on several determinants of children's fruit and vegetable intake. Based on the EnRG framework, other literature and the aims of the Learning Street, five relevant determinants are selected: (i) knowledge; (ii) taste preferences; (iii) intention; (iv) skills; and (v) attitude.

Using child-reported questionnaires, the present study aims to answer the following key questions:

What are the short-term and longer-term effects of the Kokkerelli Learning Street on children's:

* Knowledge regarding fruit and vegetable consumption?
* Intentions regarding fruit and vegetable consumption?
* Attitude regarding fruit and vegetable consumption?
* Liking of fruit and vegetables?
* Skills regarding fruit and vegetable preparation?
* Fruit and vegetable intake?

ELIGIBILITY:
Inclusion Criteria:

* Student of study years five to eight of one of the predetermined primary schools

Exclusion Criteria:

* School classes who already participated in the Kokkerelli Learning Street during previous school years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla Hahnraths, MSc, Principal Investigator — PhD candidate
Locations (1):
- Kids University for Cooking, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
It is not our intention to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were children in study years five and six (internationally comparable to grades three and four; aged 8-10 years) from primary schools in Northern Limburg, the Netherlands. Researchers and employees of Kids University for Cooking informed the children and parents about the study both orally and via information brochures (containing information about the study's purpose, procedures, and data handling). Informed consent was obtained from all parents of the participating children.
Groups:
- Intervention Group: The classes included in this group participate in the Kokkerelli Learning Street; a school-based nutrition education programme included classroom-based lessons, a visit to a grower's farm and a cooking workshop.
  Kokkerelli Learning Street: The Kokkerelli Learning Street focusses on one specific food product (kale, tomato, asparagus, pepper, strawberry, blue berry, mushroom, carrot, or leek) and consists of multiple components:
  1. An introduction lesson at school. Children are introduced to the product and familiarised with growing and harvesting processes and the importance of the product regarding health.
  2. A visit to a grower's farm during which children are introduced to the precise planting, growing and harvesting procedures of the product. Children are allowed to enter the facilities (e.g., the greenhouse) and observe and experience the farming of the product.
  3. A cooking workshop at the facilities of Kids University for Cooking BV. Children prepare a meal with help of volunteers. After preparing the meal, children help to set the table and consume their self-prepared meal.
  4. An evaluation lesson at school. Children evaluate the Learning Street together with their peers and teacher.
- Control group: The school classes included in the control group were chosen from a pool of primary schools already participating in another research project on the effects of school-based health-promoting initiatives on children's health and well-being (no publications on this study are available as the study is still ongoing). From this pool, classes from schools that were not (planning on) implementing nutrition-related and/or physical activity (PA)-related health-promoting initiatives in the context of this project were eligible to be included in the control group of the present study.
Period: Overall Study
Arm/Group | Intervention Group | Control group
Started | 61 | 165
Completed | 60 | 132
Not Completed | 1 | 33
Not completed — Not meeting criteria for data analysis | 1 | 15
Not completed — Administrative error | 0 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 60 | 132 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (0.5) | 8.6 (0.7) | 8.5 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 77 | 113
  Male | 24 | 55 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Western background (European countries (excluding Turkey), North America, Japan, Indonesia,Oceania) | 52 | 127 | 179
  Non-Western background | 8 | 5 | 13
Knowledge (mean correct) [Mean (Standard Deviation); unit: score on a scale] — The children's knowledge was assessed by six true/false questions based on the information provided in the learning street. A correct answer was scored as 1; an incorrect answer was scored as 0. A mean summary score of the number of correct answers was computed by dividing the number of correct answers by the total number of items that were answered (mean summary score could range from 0 (low knowledge) to 6 (high knowledge)).
  score on a scale | 3.0 (1.6) | 3.2 (1.2) | 3.2 (1.3)
Intention (mean score) [Mean (Standard Deviation); unit: score on a scale] — Two questions were used to assess intention, concerning participants' plans to consume or cook a meal containing the FV product, and were assessed on a five-point Likert scale from 1 = "no, I do not want to" to 5 = "yes I want to" with an additional answer option "I do not know". Mean intention was calculated by adding the scores of the questions that were answered and dividing them by the amount of answered questions (mean summary score could range from 1 (low intention) to 5 (high intention)).
  score on a scale | 3.9 (1.1) | 3.1 (1.3) | 3.4 (1.3)
Taste preferences (mean score) [Mean (Standard Deviation); unit: score on a scale] — Three questions were developed regarding taste preferences (e.g., "What do you think about the taste of the FV product?") (five-point Likert scale from 1 = "I do not like it" to 5 = "I like it very much", with an additional answer option "never tried"). Mean taste preferences were calculated by adding the scores of the questions that were answered and dividing them by the amount of answered questions (mean summary score could range from 1 (low taste preferences) to 5 (high taste preferences)).
  score on a scale | 3.6 (1.1) | 3.5 (1.2) | 3.5 (1.2)
Attitude towards addressed FV product (mean score) [Mean (Standard Deviation); unit: score on a scale] — Two questions and scales for attitude ("How much do you think the target behaviors are clever, interesting, nice, cool, and tasty?") were used as described by Ajzen and Fishbein and previously used in comparable research. From these questions, a mean summary score for (1 attitude towards FV product assessed in questionnaire and (2 general attitude towards healthy products were calculated by adding scores of the answered questions and dividing them by the amount of answered questions. For both attitude scores, mean summary score could range from 1 (negative attitude) to 5 (positive attitude).
  score on a scale | 2.7 (0.9) | 2.6 (0.9) | 2.6 (0.9)
General attitude towards healthy food (mean score) [Mean (Standard Deviation); unit: score on a scale] — Two questions and scales for attitude ("How much do you think the target behaviors are clever, interesting, nice, cool, and tasty?") were used as described by Ajzen and Fishbein and previously used in comparable research. From these questions, a mean summary score for (1 attitude towards FV product assessed in questionnaire and (2 general attitude towards healthy products were calculated by adding scores of the answered questions and dividing them by the amount of answered questions. For both attitude scores, mean summary score could range from 1 (negative attitude) to 5 (positive attitude).
  score on a scale | 3.0 (0.9) | 3.1 (0.9) | 3.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Fruit and Vegetable Knowledge at 3 Months After the Evaluation Lesson
Description: Knowledge will be assessed by six knowledge questions in the child questionnaire. A total knowledge score based on the number of correct answers will be calculated. The minimum score that can be obtained is 0, indicating low knowledge. The maximum score that can be obtained is 6, indicating high knowledge.
Time Frame: Baseline, directly after the evaluation lesson (approximately three weeks after baseline), three months after the evaluation lesson
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control group
Number analyzed (Participants) | 60 | 132
score on a scale
  T1 (directly after intervention, approximately three weeks after baseline) | 4.1 (1.09) | 3.5 (1.33)
  T2 (three months after intervention) | 3.7 (1.31) | 3.6 (1.24)
Statistical Analysis 1: Comparison: Control group; Statistical analysis at T1 (directly after the evaluation lesson); Test type: Other; p = 0.001, Regression, Linear; A three-level linear mixed model analysis, with classes as third level, participants as second level, and measurements as first level, was used
Statistical Analysis 2: Comparison: Control group; Statistical analysis at T2 (three months after the evaluation lesson); Test type: Other; p = 0.31, Regression, Linear; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline Intention to Consume Fruit and Vegetables at Three Months After the Evaluation Lesson
Description: Questions assessing intention will concern participants' plans to consume or cook a meal containing the specific food product in the future and will be assessed on a scale from 1='I don't know' to 6='yes I will'. A mean score will be calculated to assess intention. The minimum score that can be obtained is 0, indicating low intention. The maximum score that can be obtained is 6, indicating high intention.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control group
Number analyzed (Participants) | 60 | 132
score on a scale
  T1 (directly after intervention, approximately three weeks after baseline) | 4.1 (0.91) | 3.2 (1.25)
  T2 (three months after intervention) | 3.8 (1.28) | 3.3 (1.44)
Statistical Analysis 1: Comparison: Control group; Statistical analysis at T1 (directly after evaluation lesson); Test type: Other; p = 0.55, Regression, Linear; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control group; Statistical analysis at T2 (three months after evaluation lesson); Test type: Other; p = 0.33, Regression, Linear; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline Attitude Towards Fruit and Vegetable (Consumption) at 3 Months After the Evaluation Lesson
Description: Questions for attitude ('How much do you think the target behaviours are clever/interesting and nice/cool/tasty?') will be used as described by Ajzen and Fishbein and as previously used in comparable research. They will have response options ranging from 1='no, not at all' to 5='yes, totally'. A mean score will be calculated to assess attitude.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control group
Number analyzed (Participants) | 60 | 132
score on a scale
  T1 (directly after the intervention, approximately three weeks after baseline) | 2.8 (0.97) | 2.3 (0.89)
  T2 (three months after the intervention) | 2.6 (0.96) | 2.4 (0.93)
Statistical Analysis 1: Comparison: Control group; Statistical analysis at T1 (directly after evaluation lesson); Test type: Other; p = 0.004, Regression, Linear; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control group; Statistical analysis at T2 (three months after evaluation lesson); Test type: Other; p = 0.84, Regression, Linear; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Change From Baseline Taste Preferences for Fruit and Vegetables at 3 Months After the Evaluation Lesson
Description: Three questions will be used for taste preferences (e.g., 'What do you think about the taste of the food product?') (scale from 1='never tried' to 6='I like it very much'). A mean score will be calculated to assess taste preferences.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control group
Number analyzed (Participants) | 60 | 132
score on a scale
  T1 (directly after the intervention, approximately three weeks after baseline) | 3.8 (1.08) | 3.4 (1.18)
  T2 (three months after the intervention) | 3.7 (1.06) | 3.4 (1.21)
Statistical Analysis 1: Comparison: Control group; Statistical analysis at T1 (directly after evaluation lesson); Test type: Other; p = 0.002, Regression, Linear; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control group; Statistical analysis at T2 (three months after evaluation lesson); Test type: Other; p = 0.16, Regression, Linear; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Change From Baseline Attitude Towards Healthy Food Products at 3 Months After the Evaluation Lesson
Description: Questions for attitude ('How much do you think the target behaviours are clever, interesting, nice, cool, and tasty?') will be used as described by Ajzen and Fishbein and as previously used in comparable research. They will have response options ranging from 1='no, not at all' to 5='yes, totally'. A mean score will be calculated to assess attitude.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control group
Number analyzed (Participants) | 60 | 132
score on a scale
  T1 (directly after the intervention, approximately three weeks after baseline) | 3.0 (0.93) | 2.8 (0.97)
  T2 (three months after the intervention) | 2.9 (1.05) | 2.8 (0.89)
Statistical Analysis 1: Comparison: Control group; Statistical analysis at T1 (directly after evaluation lesson); Test type: Other; p = 0.01, Regression, Linear; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control group; Statistical analysis at T2 (three months after evaluation lesson); Test type: Other; p = 0.19, Regression, Linear; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse effects were monitored at three time points: Baseline, directly after the evaluation lesson (approximately three weeks after baseline), three months after the evaluation lesson.
Arm/Group | Intervention Group | Control group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/165
Other Adverse Events (participants affected / at risk) | 0/61 | 0/165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04190680/Prot_SAP_ICF_000.pdf